CLINICAL TRIAL: NCT03401541
Title: Pilot Clinical Trial to Evaluate the Pharmacokinetics of Orally Administered 25-hydroxyvitamin D3 and Vitamin D3 in Healthy Adults and Adults With a History of Intestinal Malabsorption
Brief Title: 25-Hydroxyvitamin D Pharmacokinetic Study
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Boston University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: H-37167
Record Dates: First submitted 2018-01-10; First posted 2018-01-17 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-06

CONDITIONS: Vitamin D Deficiency; Fat Malabsorption
Keywords: Calcifediol (25(OH)D); Calciferol (Vitamin D)
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Calcifediol; Cholecalciferol; Vitamin D

STUDY DESIGN:
Intervention Model Description: Each arm will first receive 25(OH)D and then vitamin D or vitamin D and then 25(OH)D
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Fat-Mal, calcifediol then calciferol (Experimental): Participants with diagnosed fat malabsorption syndrome will initially receive one capsule of calcifediol for the first round of blood draws and then receive one capsule of calciferol for the second round.
  Interventions: Drug: Calcifediol; Drug: Calciferol
- Fat-Mal, calciferol then calcifediol (Experimental): Participants with diagnosed fat malabsorption syndrome will initially receive one capsule of calciferol for the first round of blood draws and then receive one capsule of calcifediol for the second round.
  Interventions: Drug: Calcifediol; Drug: Calciferol
- Non Fat-Mal, calcifediol then calciferol (Experimental): Participants that do not have a diagnosed fat malabsorption syndrome will initially receive one capsule of calcifediol for the first round of blood draws and thenreceive one capsule of calciferol for the second round.
  Interventions: Drug: Calcifediol; Drug: Calciferol
- Non Fat-Mal, calciferol then calcifediol (Experimental): Participants that do not have a diagnosed fat malabsorption syndrome will initially receive one capsule of calciferol for the first round of blood draws and then receive one capsule of calcifediol for the second round.
  Interventions: Drug: Calcifediol; Drug: Calciferol

INTERVENTIONS:
Drug: Calcifediol — One capsule of 900 micrograms of 25(OH)D
  Other Names: 25(OH)D
Drug: Calciferol — One capsule of 900 micrograms of Vitamin D
  Other Names: Vitamin D

SUMMARY:
To evaluate the pharmacokinetic parameters of orally administered 25-hydroxyvitamin D3 [25(OH)D3] and vitamin D3 from the corresponding serum concentration-time curves in healthy adults and adults with a history of intestinal malabsorption.

DETAILED DESCRIPTION:
Patients with a history of intestinal malabsorption (n=10) and healthy volunteers (n=10); (of both sexes and all ethnicities) will be recruited in this randomized double-blind crossover study. All subjects will be prescreened for 25(OH)D levels to include subjects with 25(OH)D<30 ng/ml. The subjects will be randomized to receive a single oral dose of 900 µg of either vitamin D3 or 25(OH)D3. Blood samples will be taken at baseline and at 2,4,6,8,12 hours and days 1,2,3, 7 and 14. After a washout period of at least 14 days (2 weeks) the subjects will receive in a double blinded manner a single oral dose of 900 µg of either 25(OH)D3 or vitamin D3 (depending on which one they took in the randomization) any time after the washout. Blood samples will be taken at baseline and at 2,4,6,8,12 hours and days 1,2,3,7, 14.

Serum levels of calcium, phosphorus, albumin, creatinine, intact parathyroid hormone (iPTH) will be obtained at baseline and at day 14 (or within a reasonable time if unable to come in on the exact day). Vitamin D and 25(OH)D will be determined on all the blood samples collected at the various times.

ELIGIBILITY:
Inclusion Criteria:

* Adult male or female with history of intestinal fat-malabsorption with confirmed diagnosis
* Taking vitamin D (ergocalciferol or cholecalciferol). Subjects taking vitamin D supplement of more than 2000 IUs (50 micrograms)/day) that may interfere with study endpoints must be willing and able to discontinue use of these supplements for the duration of the study and allow for at least a 14-day washout prior to prescreening and enrollment.
* Women of child bearing potential must be on birth control and not pregnant based on a negative pregnancy test at baseline for each of the 2 pharmacokinetic studies.
* Serum total 25(OH)D < 30 ng/mL

Exclusion Criteria:

* Unwilling to discontinue use of supplemental dose of vitamin D2 (ergocalciferol) or vitamin D3 (cholecalciferol) daily equivalent (2,000 IU/50 μg) 1 week or less prior to randomization and during the study
* On medications that can affect vitamin D metabolism including steroids such as prednisone, anti-seizure medications and medications to treat HIV.
* Tanning in a tanning bed at least one week before the study and throughout the duration of this study.
* Anyone anticipating going on holiday (where exposure to sun is imminent) 1 week before or during the entire study.
* Participation in the study or any reason which, in the opinion of the investigator makes adherence to a treatment or follow-up schedule unlikely
* History of elevated serum calcium
* Chronic hepatic or renal failure
* Subjects with a history of an adverse reaction to orally administered vitamin D.
* Inability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-11-01 (Actual)

PRIMARY OUTCOMES:
Change in Serum vitamin D status | 2 weeks after administration
  The serum vitamin D status (pg/mL) will be determined at multiple time points secondary to receiving a single dose of either calciferol or calcifediol. We will obtain 11 time points after each drug administration which will allow us to observe the fluctuation in vitamin D status after receiving the study drug.
Change in 25-Hydroxyvitamin D Status | 2 weeks after administration
  The serum 25(OH)D status (ng/mL) will be determined at multiple time points secondary to receiving a single dose of either calciferol or calcifediol. We will obtain 11 time points after each drug administration which will allow us to observe the fluctuation in 25(OH)D status after receiving the study drug.

SECONDARY OUTCOMES:
Serum Calcium Levels | Baseline and completion of each intervention period (2 weeks)
  Calcium levels will be drawn at baseline and at the end of each intervention period. This measure will allow us to ensure no change to baseline levels after receiving the study drug.
Serum Phosphorus Levels | Baseline and completion of each intervention period (2 weeks)
  Phosphorus levels will be drawn at baseline and at the end of each intervention period. This measure will allow us to ensure no change to baseline levels after receiving the study drug.
Serum Albumin Levels | Baseline and completion of each intervention period (2 weeks)
  Albumin levels will be drawn at baseline and at the end of each intervention period. This measure will allow us to ensure no change to baseline levels after receiving the study drug.
Serum Creatinine levels | Baseline and completion of each intervention period (2 weeks)
  Creatinine levels will be drawn at baseline and at the end of each intervention period. This measure will allow us to ensure no change to baseline levels after receiving the study drug.
Serum intact parathyroid hormone levels | Baseline and completion of each intervention period (2 weeks)
  iPTH levels will be drawn at baseline and at the end of each intervention period. This measure will allow us to ensure no change to baseline levels after receiving the study drug.

CONTACTS AND LOCATIONS:
Overall Officials: Michael F Holick, MD, PhD, Principal Investigator — Boston University
Locations (1):
- Solomon Carter Fuller Mental Health Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be available upon reasonable request to mfholick@bu.edu.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Beginning 9 month and ending 36 months following article publication.
Access Criteria: Investigators whose proposed use of the data has been approved by the current study principal investigators.

REFERENCES:
- [Derived] Charoenngam N, Kalajian TA, Shirvani A, Yoon GH, Desai S, McCarthy A, Apovian CM, Holick MF. A pilot-randomized, double-blind crossover trial to evaluate the pharmacokinetics of orally administered 25-hydroxyvitamin D3 and vitamin D3 in healthy adults with differing BMI and in adults with intestinal malabsorption. Am J Clin Nutr. 2021 Sep 1;114(3):1189-1199. doi: 10.1093/ajcn/nqab123. PMID 34008842